CLINICAL TRIAL: NCT00924794
Title: A Retrospective Epidemiological Study of Natural History of HPV Infections in Women Aged 18 Years and Above With Recurrent Conization Following a Primary Conization for High Grade Lesions/ Microinvasive Cervical Carcinomas, in Norway
Brief Title: Study of Natural History of Human Papillomavirus (HPV) Infections in Adult Women With Recurrent Conizations in Norway
Status: Terminated | Type: Observational
Why Stopped: This complex study included a pilot and a main part. As the results of the pilot study were satisfying and conclusive, the main study was not performed.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112674
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Infections, Papillomavirus
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort A: Women aged 18 years and above, diagnosed with high grade lesions or microinvasive cervical carcinomas in primary conization performed and registered in the Cancer Registry of Norway, and presenting with recurrent conization with high grade lesions or microinvasive cervical carcinoma or invasive cervical carcinoma.
  Interventions: Procedure: Cancer Registry of Norway (database)

INTERVENTIONS:
Procedure: Cancer Registry of Norway (database) — Review of database to identify women with primary conization presenting with high grade lesions/ microinvasive cervical carcinomas. Recurrent cones with high grade lesions/ microinvasive cervical carcinomas or invasive cervical cancer will be identified for all women with primary cones.

SUMMARY:
This is a register-based, epidemiological study of HPV type distribution in women aged 18 years and above with recurrent conization following a primary conization for high grade lesions/ microinvasive carcinomas. This study will involve data collection from different databases in the Cancer Registry of Norway.

DETAILED DESCRIPTION:
This protocol posting has been updated following Protocol Amendment 1 (02 April 2010). The sections impacted are: enrolment, outcome measures and eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

All subjects must meet the following criteria at study entry:

* Women aged 18 years and above at the time of the collection of the primary cone specimen;
* Who have undergone for the first time a conization due to high grade lesions or microinvasive cervical carcinomas, histologically diagnosed in 2003, with possible extension backwards in time;
* Availability of recurrent cone specimen with high grade lesions/ microinvasive cervical carcinomas or invasive cervical cancer;
* Availability in designated local laboratories of the primary and recurrent cone specimens;
* The cone specimen was adequately preserved;
* Written informed consent obtained from the subject. If the subject is deceased, the cone and biopsy specimens will be used according to prior approval from the Ethics Committee.

Exclusion Criteria:

None.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 18 years and above registered in the Cancer Registry of Norway.
Sampling Method: Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
HPV-types as single group considered as new infections in recurrent conizations with high grade lesions, microinvasive cervical carcinomas or ICC diagnosis. | At the end of the study.
HPV-types as single group considered as persistent infections in recurrent conizations with high grade lesions, microinvasive cervical carcinomas or ICC diagnosis. | At the end of the study.

SECONDARY OUTCOMES:
HPV-types as individual types or as different groups considered as new infections in recurrent conizations presenting high grade lesions, microinvasive cervical carcinomas or ICC diagnosis. | At the end of the study.
HPV-types as individual types or as different groups considered as persistent infections in recurrent conizations presenting high grade lesions, microinvasive cervical carcinomas or ICC diagnosis. | At the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bergen, Norway

REFERENCES:
- [Derived] Vintermyr OK, Iversen O, Thoresen S, Quint W, Molijn A, de Souza S, Rosillon D, Holl K. Recurrent high-grade cervical lesion after primary conization is associated with persistent human papillomavirus infection in Norway. Gynecol Oncol. 2014 May;133(2):159-66. doi: 10.1016/j.ygyno.2014.03.004. Epub 2014 Mar 11. PMID 24631451